CLINICAL TRIAL: NCT01083420
Title: The Efficacy of Topical Minocycline in Managing Symptomatic Oral Lichen Planus. A Randomized Controlled Trial
Brief Title: The Efficacy of Topical Minocycline in Managing Symptomatic Oral Lichen Planus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Noam Yarom, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SHEBA-09-7335-NY-CTIL
Record Dates: First submitted 2010-03-07; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; Minocycline; Dexamethasone
MeSH Terms: conditions — Lichen Planus, Oral; cyclopia sequence | interventions — Minocycline; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone 0.01% mouthwash
  Interventions: Drug: Dexamethasone
- Minocycline (Experimental): Minocycline 0.2% mouthwash
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — Minocycline 0.2% mouthwash
  Arms: Minocycline
Drug: Dexamethasone — Dexamethasone 0.01% mouthwash
  Arms: Dexamethasone

SUMMARY:
The aim of the present study is to assess the clinical efficacy of topical minocyclin in managing of symptoms associated with oral lichen planus (OLP). The rationale of the study is based on our previous studies demonstrating the beneficial effect of minocyclin mouthwash on recurrent aphthous stomatitis. The planned study will be a randomized controlled, cross-over trail. Patients with symptomatic OLP will randomly receive minocycline or dexamethasone rinses.

The patients will rinse and expectorate 5 ml of the 1st mouthwash 4 times daily for 14 days. Subjects will complete a daily follow-up form that includes data regarding the daily intensity of pain (using VAS) caused by OLP and regarding possible side effects. After a washout period (at least 14 days) the patients will repeat the protocol with the second mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* OLP patients (Biopsy proven)

Exclusion Criteria:

* Known allergy to Dexamethasone or Minocycline
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2011-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
symptoms relief | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noam Yarom, DMD, Principal Investigator — Sheba Medical Center